CLINICAL TRIAL: NCT00375076
Title: Prevention of Venous Thrombosis in Cancer Patients: A Prospective, Randomized, Double-blind Study Comparing Two Different Dosages of Low-molecular Weight Heparin
Brief Title: Comparison of Two Different Dosages of Low-molecular Weight Heparin in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Sabine Eichinger, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ODEXA1
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Enoxaparin

INTERVENTIONS:
Drug: enoxaparin

SUMMARY:
In a prospective, randomized, double-blind trial, the effects of two different dosages of LMWH (5000 anti-Xa U od sc and 10 000 anti-Xa U od sc daily) on markers of hemostatic system and thrombin generation will be investigated in non-surgical cancer patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Patients (> 18 years) with active cancer and at least one of the following indications for thromboprophylaxis with LMWH:

* Immobilization
* History of VTE
* Acute inflammation
* Heart failure (NYHA class III or IV)
* Respiratory failure

Exclusion Criteria:

* Indication for LMWH or UFH at therapeutic dosages
* Treatment with antithrombotics (vitamin K antagonists, acetylsalicylic acid, clopidogrel) for reasons other than prevention of VTE (e.g. atrial fibrillation, myocardial infarction)
* Contraindication for the treatment with LMWH
* Major surgery within the last 4 weeks; minor surgery within the last week
* Thrombocytopenia (< 100.000/μl)
* Prolonged prothrombin time
* Prolonged activated partial thromboplastin time (aPTT)
* History of heparin-induced thrombocytopenia
* Bodyweight < 50 kg or > 100 kg
* Renal insufficiency (creatinine > 2 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Eichinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria